CLINICAL TRIAL: NCT03895450
Title: Improving Symptom Burden in Individuals With Persistent Post Concussive Symptoms: A Step-wise Aerobic Exercise Trial
Brief Title: Treating Persistent Post-concussion Symptoms With Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Hotchkiss Brain Institute, University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: REB18-1329
Record Dates: First submitted 2019-02-11; First posted 2019-03-29 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Brain Injuries, Traumatic; Concussion, Brain; Mild Traumatic Brain Injury; Post-Concussion Syndrome
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Post-Concussion Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Allocation will be concealed through the use of sequentially numbered, opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Protocol (AEP) (Experimental): Symptom threshold will be determined at baseline and repeated every 3 weeks using the Buffalo Concussion Treadmill Test. Briefly, there will be an initial 4min warm up at 1.7mph. The protocol will start with treadmill speed se to 3.3 mph and 0.0% incline. Each subsequent minute, the incline will increase by 1.0% to a max of 15%. At 15% grade, if the participant is still able to continue, treadmill speed will increase by 0.4mph each minute. Heart rate (HR) and rating of perceived excretion (RPE Borg scale) will be measured every minute. The test will be terminated upon symptom exacerbation at which time HR and RPE will be recorded. Every 3 weeks the symptom threshold test will be repeated for all participants and exercise prescription will be adjusted accordingly.
  Interventions: Behavioral: Aerobic Exercise Protocol
- Stretching Protocol (SP) (Placebo Comparator): The exercise testing for the stretching protocol to determine exercise prescription will be the same as described above.
  Interventions: Behavioral: Aerobic Exercise Protocol; Behavioral: Stretching Protocol

INTERVENTIONS:
Behavioral: Aerobic Exercise Protocol — Participants randomized to AEP will be asked to exercise 30 minutes per day or until symptom exacerbation, 5 days per week either at home, outdoors or at a fitness facility of choice. The assigned exercise prescription target will be 70-80% of the maximum HR achieved during the treadmill test. HR monitors will be provided to monitor exercise intensity.
Behavioral: Stretching Protocol — Participants will follow a stretching protocol for 30 minutes a day, 5 days a week. Individuals in the SP group will be given a booklet explaining a low-impact breathing and stretching program developed at the University of Buffalo. All stretches will explained and demonstrated by a member of the study team prior to commencement of the program. Stretches focus on lower extremity muscles. During the protocol HR should be low as to not exceed 50% of age predicted max. A HR monitor will be worn during stretching.
  Arms: Stretching Protocol (SP)

SUMMARY:
The objective of this study is to investigate an aerobic exercise program as a treatment for adults with persistent post-concussive symptoms (PPCS) following mild traumatic brain injury. In this delayed-start trial participants will be initially randomized into either a 6-week low-impact stretching protocol or 12-week aerobic exercise protocol. Following the completion of the stretching protocol participants will continue on to complete the aerobic exercise protocol in full. 56 participants aged 18-65 yrs will be recruited from the Calgary Brain Injury Program (CBIP), including the Early Concussion Education Program at Foothills Medical Centre, Calgary Pain Program, University of Calgary Sports Medicine Centre acute concussion clinic and a physiotherapy clinic (Tower Physio) all of which are located in Calgary, Alberta, Canada. Participants will complete an online follow up (symptom questionnaires and questions regarding exercise behaviour) 3 and 9 weeks post intervention.

DETAILED DESCRIPTION:
Demographic information will be collected prior to study participation and include age, sex, education, family medical history, past medical history, concussion history, litigious status and medication use. The PAR-Q+ questionnaire will be completed to determine readiness for exercise by a physician. Baseline questionnaires will be completed, such as the Fatigue Severity Scale (FSS), Generalized Anxiety Disorder Scale (GAD-7), Headache Intensity Scale-6 (HIT-6), Patient Health Questionnaire(PHQ-9), Epworth Sleepiness Scale(ESS) and Quality of Life After Brain Injury(QOLIBRI), Rivermead Post Concussion Symptoms Questionnaire (RPQ), Modified Godin Leisure-Time Exercise Questionnaire(GLTQ), Rapid Assessment Disuse Index (RADI) and Postconcusion Syndrome Checklist (PCSC). Pre- and post-intervention blood samples will be collected from all participants. Participants will be asked to perform a tactile assessment pre- and post-intervention. Sleep will be monitored using wrist-based actigraphy and a sleep diary for 3-6 days/nights prior to the intervention start and for five days following completion of the exercise protocol. Pre and post magnetic resonance spectroscopy (MRS) will also be completed. Participants will be randomized to a structured aerobic exercise protocol (AEP) or stretching protocol, followed by aerobic exercise protocol(SP+AEP) with a random number generator. Both groups will undergo exercise testing using the Buffalo Concussion Treadmill Test to determine exercise prescription. Upon completion of SP, participants will continue on to the AEP and complete it in full. Following the exercise protocols, all questionnaires will be completed post-intervention. At 3 and 9 weeks following protocol completion, online follow surveys will be completed to assess symptom burden (RPQ, QOLIBRI, HIT-6, ESS, FSS) along with questions regarding current exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild traumatic brain injury (mTBI) based on the American Congress of Rehabilitation Medicine (ACRM) criteria.
* mTBI occurrence from 3 months to 5 years from study start date
* Diagnosis of persistent post-concussion symptoms based on the ICD-10 criteria.
* Cleared for physical activity based on The Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) by treating physician
* exercise intolerance (inability to exercise at pre-injury intensity/duration due to acute presentation of symptoms)

Exclusion Criteria:

* past medical history of neurological disorders (i.e., Parkinson's disease, neuromuscular disorders)
* contraindications to MRI
* cardiopulmonary disorder
* chronic musculoskeletal condition
* psychiatric disorder other than depression and/or anxiety (i.e., schizophrenia, bipolar disorder)
* cancer
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Change in symptom burden | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP, 3-weeks post-AEP, 9-weeks post-AEP
  Rivermead Post-concussion Symptoms Questionnaire (RPQ): an instrument developed to assess the frequency and severity of 16 common post-concussion symptoms. On this paper and pencil tool, patients rate the extent to which their symptoms (compared to their pre-injury levels) have become more problematic over the past 24 hours using a rating scale from 0-4 (0=not experienced, 1=no more of a problem, 2=mild problem, 3=moderate problem, 4=severe problem). A total symptom score is calculated out of 64.

SECONDARY OUTCOMES:
Change in sleep duration | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  Wrist actigraphy confirmed by a sleep diary. An actigraph (MotionWatch8 [CamNTech]) watch will be worn on the non-dominant wrist during nighttime hours. Actigraphy results will be confirmed by a sleep diary completed in the morning.
Change in daytime sleepiness | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP, 3-weeks post-AEP, 9-weeks post-AEP
  Epworth Sleepiness Scale (ESS): measure of daytime sleepiness. This scale rates the chance of dozing off on a scale of 0-3 (0= would never doze, 1= slight chance of dozing, 2= moderate chance of dozing, 3=high chance of dozing) in 8 different situations.
Change in blood derived neurotrophic factor (BDNF) | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  BDNF: serum BDNF, a neurotropic factor involved in neuronal repair after injury, will be analyzed for change in serum concentration
Change in cytokine profile | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  Cytokine profile: serum levels of multiple cytokines will be used to characterise chronic inflammatory changes
Change in telomere length (TL) | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  Telomeres are non-coding sequences of DNA that are found at the end of linear eukaryotic chromosomes thought to play a role in DNA strand repair. TL length will be analyzed using whole blood collected across time points.
Change in fatigue | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP, 3-weeks post-AEP, 9-weeks post-AEP
  Fatigue Severity Scale (FSS): 9 instrument questionnaire. Each item is rated on a 7 point likert scale (1= Strongly disagree, 7=strongly agree). Total score is calculated by adding the score from each item producing a total out of 63. A final item asks to "Please mark "X" on a number line which describes your global fatigue with 0 being worst and 10 being normal."
Change in anxiety | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  Generalized Anxiety Disorder (GAD-7): a 7-item tool where each item is rated on frequency over a 2 week period based on a 0-3 scale (0=not at all, 1=several days, 2=more than half the days, 3=nearly every day). The total score ranges from 0 to 21, with scores indicating severity of anxiety (ie. 0-5= mild, 6-10= moderate, 11-15= moderately severe, 16-21= very severe).
Change in function related to headaches | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP, 3-weeks post-AEP, 9-weeks post-AEP
  Headache Impact Test (HIT-6): a global measure of headache impact. Addresses the 6 categories of headache impact including social, ADL, and cognitive functioning, vitality, psychological distress, and severity of headache pain. Each question is scored on a 5 point scale (never, rarely, sometimes, very often, always). Total score can range from 36-78, with higher total score indicating greater impact.
Change in depression | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-weeks of AEP
  Patient Health Questionnaire-9 (PHQ-9): 9 item tool to assess the presence and severity of depressive symptoms. Each item is rated based on the frequency of occurrence in the past 2 weeks and is graded ona 0-3 scale (0=not at all, 1=several days, 2= more than half of the days, 3= nearly every day). A stand-alone question asks to rate how difficult problems have made completing tasks at home, doing work, and getting along with people. This is graded on a 4-point scale from not difficult at all to extremely difficult. Total score is calculated out of 27, with the value indicating severity of depression (ie. 0-4= none to mild, 5-9= mild, 10-14= moderate, 15-19= moderately severe, and 20-27= very severe).
MRS quantification of GABA/Glutathione | Repeated measure: Pre-intervention, after 6-weeks of SP/AEP, after 12-week of AEP
  Changes in GABA, glutathione and glutamate in the dorsolateral perefrontal cortex between AEP and SP group at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Chantel T Debert, MD MSc FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University Of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korley FK, Kelen GD, Jones CM, Diaz-Arrastia R. Emergency Department Evaluation of Traumatic Brain Injury in the United States, 2009-2010. J Head Trauma Rehabil. 2016 Nov/Dec;31(6):379-387. doi: 10.1097/HTR.0000000000000187. PMID 26360006
- [Background] Cassidy JD, Carroll LJ, Peloso PM, Borg J, von Holst H, Holm L, Kraus J, Coronado VG; WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. Incidence, risk factors and prevention of mild traumatic brain injury: results of the WHO Collaborating Centre Task Force on Mild Traumatic Brain Injury. J Rehabil Med. 2004 Feb;(43 Suppl):28-60. doi: 10.1080/16501960410023732. PMID 15083870
- [Background] Coenen M, Cabello M, Umlauf S, Ayuso-Mateos JL, Anczewska M, Tourunen J, Leonardi M, Cieza A; PARADISE Consortium. Psychosocial difficulties from the perspective of persons with neuropsychiatric disorders. Disabil Rehabil. 2016;38(12):1134-45. doi: 10.3109/09638288.2015.1074729. Epub 2015 Aug 18. PMID 26289372
- [Background] Olesen J, Leonardi M. The burden of brain diseases in Europe. Eur J Neurol. 2003 Sep;10(5):471-7. doi: 10.1046/j.1468-1331.2003.00682.x. PMID 12940825
- [Background] Humphreys I, Wood RL, Phillips CJ, Macey S. The costs of traumatic brain injury: a literature review. Clinicoecon Outcomes Res. 2013 Jun 26;5:281-7. doi: 10.2147/CEOR.S44625. Print 2013. PMID 23836998
- [Background] Lange RT, Brickell TA, Kennedy JE, Bailie JM, Sills C, Asmussen S, Amador R, Dilay A, Ivins B, French LM. Factors influencing postconcussion and posttraumatic stress symptom reporting following military-related concurrent polytrauma and traumatic brain injury. Arch Clin Neuropsychol. 2014 Jun;29(4):329-47. doi: 10.1093/arclin/acu013. Epub 2014 Apr 9. PMID 24723461
- [Background] Waljas M, Iverson GL, Lange RT, Liimatainen S, Hartikainen KM, Dastidar P, Soimakallio S, Ohman J. Return to work following mild traumatic brain injury. J Head Trauma Rehabil. 2014 Sep-Oct;29(5):443-50. doi: 10.1097/HTR.0000000000000002. PMID 24263178
- [Background] Lange RT, Iverson GL, Rose A. Depression strongly influences postconcussion symptom reporting following mild traumatic brain injury. J Head Trauma Rehabil. 2011 Mar-Apr;26(2):127-37. doi: 10.1097/HTR.0b013e3181e4622a. PMID 20631632
- [Background] Mychasiuk R, Hehar H, Ma I, Candy S, Esser MJ. Reducing the time interval between concussion and voluntary exercise restores motor impairment, short-term memory, and alterations to gene expression. Eur J Neurosci. 2016 Oct;44(7):2407-2417. doi: 10.1111/ejn.13360. Epub 2016 Aug 31. PMID 27521273
- [Background] Hearing CM, Chang WC, Szuhany KL, Deckersbach T, Nierenberg AA, Sylvia LG. Physical Exercise for Treatment of Mood Disorders: A Critical Review. Curr Behav Neurosci Rep. 2016 Dec;3(4):350-359. doi: 10.1007/s40473-016-0089-y. Epub 2016 Oct 14. PMID 28503402
- [Background] Stroth S, Hille K, Spitzer M, Reinhardt R. Aerobic endurance exercise benefits memory and affect in young adults. Neuropsychol Rehabil. 2009 Apr;19(2):223-43. doi: 10.1080/09602010802091183. Epub 2008 Jun 1. PMID 18609015
- [Background] Geneen LJ, Moore RA, Clarke C, Martin D, Colvin LA, Smith BH. Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews. Cochrane Database Syst Rev. 2017 Apr 24;4(4):CD011279. doi: 10.1002/14651858.CD011279.pub3. PMID 28436583
- [Background] Larun L, Brurberg KG, Odgaard-Jensen J, Price JR. Exercise therapy for chronic fatigue syndrome. Cochrane Database Syst Rev. 2017 Apr 25;4(4):CD003200. doi: 10.1002/14651858.CD003200.pub7. PMID 28444695
- [Background] Gurley JM, Hujsak BD, Kelly JL. Vestibular rehabilitation following mild traumatic brain injury. NeuroRehabilitation. 2013;32(3):519-28. doi: 10.3233/NRE-130874. PMID 23648606
- [Background] Zhang QW, Deng XX, Sun X, Xu JX, Sun FY. Exercise promotes axon regeneration of newborn striatonigral and corticonigral projection neurons in rats after ischemic stroke. PLoS One. 2013 Nov 19;8(11):e80139. doi: 10.1371/journal.pone.0080139. eCollection 2013. PMID 24260348
- [Background] Piao CS, Stoica BA, Wu J, Sabirzhanov B, Zhao Z, Cabatbat R, Loane DJ, Faden AI. Late exercise reduces neuroinflammation and cognitive dysfunction after traumatic brain injury. Neurobiol Dis. 2013 Jun;54:252-63. doi: 10.1016/j.nbd.2012.12.017. Epub 2013 Jan 8. PMID 23313314
- [Background] Molteni R, Zheng JQ, Ying Z, Gomez-Pinilla F, Twiss JL. Voluntary exercise increases axonal regeneration from sensory neurons. Proc Natl Acad Sci U S A. 2004 Jun 1;101(22):8473-8. doi: 10.1073/pnas.0401443101. Epub 2004 May 24. PMID 15159540
- [Background] Cotman CW, Berchtold NC, Christie LA. Exercise builds brain health: key roles of growth factor cascades and inflammation. Trends Neurosci. 2007 Sep;30(9):464-72. doi: 10.1016/j.tins.2007.06.011. Epub 2007 Aug 31. PMID 17765329
- [Background] Griesbach GS, Hovda DA, Gomez-Pinilla F. Exercise-induced improvement in cognitive performance after traumatic brain injury in rats is dependent on BDNF activation. Brain Res. 2009 Sep 8;1288:105-15. doi: 10.1016/j.brainres.2009.06.045. Epub 2009 Jun 23. PMID 19555673
- [Background] Fogelman D, Zafonte R. Exercise to enhance neurocognitive function after traumatic brain injury. PM R. 2012 Nov;4(11):908-13. doi: 10.1016/j.pmrj.2012.09.028. PMID 23174558
- [Background] Wogensen E, Mala H, Mogensen J. The Effects of Exercise on Cognitive Recovery after Acquired Brain Injury in Animal Models: A Systematic Review. Neural Plast. 2015;2015:830871. doi: 10.1155/2015/830871. Epub 2015 Oct 5. PMID 26509085
- [Background] Martinsen S, Flodin P, Berrebi J, Lofgren M, Bileviciute-Ljungar I, Mannerkorpi K, Ingvar M, Fransson P, Kosek E. The role of long-term physical exercise on performance and brain activation during the Stroop colour word task in fibromyalgia patients. Clin Physiol Funct Imaging. 2018 May;38(3):508-516. doi: 10.1111/cpf.12449. Epub 2017 Jun 18. PMID 28627125
- [Background] Edwards T, Pilutti LA. The effect of exercise training in adults with multiple sclerosis with severe mobility disability: A systematic review and future research directions. Mult Scler Relat Disord. 2017 Aug;16:31-39. doi: 10.1016/j.msard.2017.06.003. Epub 2017 Jun 12. PMID 28755682
- [Background] Clark PJ, Brzezinska WJ, Thomas MW, Ryzhenko NA, Toshkov SA, Rhodes JS. Intact neurogenesis is required for benefits of exercise on spatial memory but not motor performance or contextual fear conditioning in C57BL/6J mice. Neuroscience. 2008 Sep 9;155(4):1048-58. doi: 10.1016/j.neuroscience.2008.06.051. Epub 2008 Jul 1. PMID 18664375
- [Background] Erickson KI, Voss MW, Prakash RS, Basak C, Szabo A, Chaddock L, Kim JS, Heo S, Alves H, White SM, Wojcicki TR, Mailey E, Vieira VJ, Martin SA, Pence BD, Woods JA, McAuley E, Kramer AF. Exercise training increases size of hippocampus and improves memory. Proc Natl Acad Sci U S A. 2011 Feb 15;108(7):3017-22. doi: 10.1073/pnas.1015950108. Epub 2011 Jan 31. PMID 21282661
- [Background] Biedermann SV, Fuss J, Steinle J, Auer MK, Dormann C, Falfan-Melgoza C, Ende G, Gass P, Weber-Fahr W. The hippocampus and exercise: histological correlates of MR-detected volume changes. Brain Struct Funct. 2016 Apr;221(3):1353-63. doi: 10.1007/s00429-014-0976-5. Epub 2014 Dec 31. PMID 25550000
- [Background] Chaddock L, Erickson KI, Prakash RS, Kim JS, Voss MW, Vanpatter M, Pontifex MB, Raine LB, Konkel A, Hillman CH, Cohen NJ, Kramer AF. A neuroimaging investigation of the association between aerobic fitness, hippocampal volume, and memory performance in preadolescent children. Brain Res. 2010 Oct 28;1358:172-83. doi: 10.1016/j.brainres.2010.08.049. Epub 2010 Aug 22. PMID 20735996
- [Background] Hehar H, Mychasiuk R. The use of telomere length as a predictive biomarker for injury prognosis in juvenile rats following a concussion/mild traumatic brain injury. Neurobiol Dis. 2016 Mar;87:11-8. doi: 10.1016/j.nbd.2015.12.007. Epub 2015 Dec 17. PMID 26709201
- [Background] Leddy J, Baker JG, Haider MN, Hinds A, Willer B. A Physiological Approach to Prolonged Recovery From Sport-Related Concussion. J Athl Train. 2017 Mar;52(3):299-308. doi: 10.4085/1062-6050-51.11.08. PMID 28387557
- [Background] Leckie RL, Oberlin LE, Voss MW, Prakash RS, Szabo-Reed A, Chaddock-Heyman L, Phillips SM, Gothe NP, Mailey E, Vieira-Potter VJ, Martin SA, Pence BD, Lin M, Parasuraman R, Greenwood PM, Fryxell KJ, Woods JA, McAuley E, Kramer AF, Erickson KI. BDNF mediates improvements in executive function following a 1-year exercise intervention. Front Hum Neurosci. 2014 Dec 11;8:985. doi: 10.3389/fnhum.2014.00985. eCollection 2014. PMID 25566019
- [Background] Merritt VC, Arnett PA. Apolipoprotein E (APOE) ϵ4 Allele Is Associated with Increased Symptom Reporting Following Sports Concussion. J Int Neuropsychol Soc. 2016 Jan;22(1):89-94. doi: 10.1017/S1355617715001022. Epub 2015 Oct 20. PMID 26483005
- [Background] Merritt VC, Rabinowitz AR, Arnett PA. The Influence of the Apolipoprotein E (APOE) Gene on Subacute Post-Concussion Neurocognitive Performance in College Athletes. Arch Clin Neuropsychol. 2018 Feb 1;33(1):36-46. doi: 10.1093/arclin/acx051. PMID 28541413
- [Background] von Steinbuechel N, Covic A, Polinder S, Kohlmann T, Cepulyte U, Poinstingl H, Backhaus J, Bakx W, Bullinger M, Christensen AL, Formisano R, Gibbons H, Hofer S, Koskinen S, Maas A, Neugebauer E, Powell J, Sarajuuri J, Sasse N, Schmidt S, Muhlan H, von Wild K, Zitnay G, Truelle JL. Assessment of Health-Related Quality of Life after TBI: Comparison of a Disease-Specific (QOLIBRI) with a Generic (SF-36) Instrument. Behav Neurol. 2016;2016:7928014. doi: 10.1155/2016/7928014. Epub 2016 Feb 1. PMID 27022207
- [Background] Esselman PC, Uomoto JM. Classification of the spectrum of mild traumatic brain injury. Brain Inj. 1995 May-Jun;9(4):417-24. doi: 10.3109/02699059509005782. PMID 7640688
- [Background] Ades PA, Grunvald MH. Cardiopulmonary exercise testing before and after conditioning in older coronary patients. Am Heart J. 1990 Sep;120(3):585-9. doi: 10.1016/0002-8703(90)90015-p. PMID 2389695
- [Background] Baker JG, Freitas MS, Leddy JJ, Kozlowski KF, Willer BS. Return to full functioning after graded exercise assessment and progressive exercise treatment of postconcussion syndrome. Rehabil Res Pract. 2012;2012:705309. doi: 10.1155/2012/705309. Epub 2012 Jan 16. PMID 22292122
- [Background] Leddy JJ, Sandhu H, Sodhi V, Baker JG, Willer B. Rehabilitation of Concussion and Post-concussion Syndrome. Sports Health. 2012 Mar;4(2):147-54. doi: 10.1177/1941738111433673. PMID 23016082
- [Background] Polak P, Leddy JJ, Dwyer MG, Willer B, Zivadinov R. Diffusion tensor imaging alterations in patients with postconcussion syndrome undergoing exercise treatment: a pilot longitudinal study. J Head Trauma Rehabil. 2015 Mar-Apr;30(2):E32-42. doi: 10.1097/HTR.0000000000000037. PMID 24721808
- [Background] Donnelly KZ, Linnea K, Grant DA, Lichtenstein J. The feasibility and impact of a yoga pilot programme on the quality-of-life of adults with acquired brain injury. Brain Inj. 2017;31(2):208-214. doi: 10.1080/02699052.2016.1225988. Epub 2016 Dec 12. PMID 27936953
- [Derived] Mercier LJ, McIntosh SJ, Boucher C, Joyce JM, Batycky J, Galarneau JM, Esser MJ, Schneider KJ, Dukelow SP, Harris AD, Debert CT. Effect of Aerobic Exercise on Symptom Burden and Quality of Life in Adults With Persisting Post-concussive Symptoms: The ACTBI Randomized Controlled Trial. Arch Phys Med Rehabil. 2025 Feb;106(2):195-205. doi: 10.1016/j.apmr.2024.10.002. Epub 2024 Oct 18. PMID 39427780
- [Derived] Mercier LJ, Fung TS, Harris AD, Dukelow SP, Debert CT. Improving symptom burden in adults with persistent post-concussive symptoms: a randomized aerobic exercise trial protocol. BMC Neurol. 2020 Feb 5;20(1):46. doi: 10.1186/s12883-020-1622-x. PMID 32024486